CLINICAL TRIAL: NCT05956522
Title: Single-center, Open, Randomized, Single-dose, Crossover Bioequivalence Study Evaluating the Use of the Subject Formulation, Empagliflozin And Linagliptin Tablets, Versus the Reference Formulation, Empagliflozin And Linagliptin Tablets (Glyxambi®), in Healthy Adult Subjects
Brief Title: Bioequivalence Study of Empagliflozin And Linagliptin Tablets in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QLG1045-01
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test/reference (Experimental): Subjects first receive a single-dose of 25 mg/5 mg test Empagliflozin And Linagliptin tablet (T, produced by Qilu Pharmaceutical (Hainan) Co., Ltd ) in the first treatment period and to receive the reference (R, Boehringer Ingelheim International GmbH & Co. KG )in the second treatment period.
  Interventions: Drug: Test Empagliflozin And Linagliptin Tablets; Drug: Reference Empagliflozin And Linagliptin tablets
- Reference/test (Experimental): Subjects first receive a single-dose of 25 mg/5 mg reference Empagliflozin And Linagliptin tablet (R, Boehringer Ingelheim International GmbH & Co. KG) in the first treatment period and to receive test tablet (T, produced by Qilu Pharmaceutical (Hainan) Co., Ltd) in the second treatment period.
  Interventions: Drug: Test Empagliflozin And Linagliptin Tablets; Drug: Reference Empagliflozin And Linagliptin tablets

INTERVENTIONS:
Drug: Test Empagliflozin And Linagliptin Tablets — specification: 25 mg/5 mg, manufacturer: Qilu Pharmaceutical (Hainan) Co., Ltd
Drug: Reference Empagliflozin And Linagliptin tablets — specification: 25 mg/5 mg, manufacturer: Boehringer Ingelheim International GmbH & Co. KG

SUMMARY:
To investigate the pharmacokinetics of the test and the reference preparation Empagliflozin And Linagliptin Tablets in healthy adult subjects by single oral administration in fasting/postprandial state, and to evaluate the bioequivalence of the two oral preparations in fasting/postprandial state.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign informed consent before the test, and fully understand the test content, process and possible adverse reactions; 2. Be able to complete the study according to the requirements of the test plan; 3. Subjects (including male subjects) agreed to have no pregnancy plan and to voluntarily take effective contraceptive measures within 3 months from the end of the study after signing the informed consent; 4. Male and female subjects aged 18 years and above; 5. Male subjects weigh at least 50kg. Female subjects weighed at least 45 kilograms. Body Mass index = weight (kg)/height 2 (m2), within the range of 19.0 to 27.0kg/m2 (including the critical value)

Exclusion Criteria:

* 1.History of specific allergies (urticaria, exfoliative dermatitis, angioedema or bronchial hypersensitivity), or allergies (e.g., allergy to two or more medications, foods such as milk and pollen), or known allergy to components of the drug or its analogues; 2. Those with a history of serious diseases such as cardiac, hepatic, renal, gastrointestinal, neurological, endocrine, respiratory and mental abnormalities, etc., which are considered inappropriate by the investigating doctor; 3. Abnormalities of clinical significance as determined by the clinician, including physical examination, vital signs, electrocardiogram or clinical laboratory tests.

  4. Previous or current history of pancreatitis; 5. Estimated glomerular filtration rate (eGFR) <90 mL/min/1.73 m2; 6. History of dysphagia or any gastrointestinal disorder that interferes with drug absorption (e.g., gastric or small bowel resection, atrophic gastritis, gastrointestinal hemorrhage, gastrointestinal bleeding); 7. Those who have difficulty in collecting blood, or cannot tolerate venipuncture, or have a history of blood or needle sickness.

  8. Female subjects who are pregnant, breastfeeding or have a positive pregnancy test result; 9. Hepatitis B surface antigen, Hepatitis C antibody, HIV antibody or syphilis antibody, any one or more of which is positive; 10. A history of substance abuse within five years, or drug use within three months prior to screening, or a positive urine drug screen.

  11. A person who has consumed an average of more than 14 units of alcohol (1 unit = 360 mL of beer or 45 mL of 40% alcohol by volume spirits or 150 mL of wine) per week during the 3 months prior to screening, or who does not agree to stop alcohol intake 24 hours prior to check-in for each cycle until the end of the cycle for which the blood sample was collected, or who has a positive breath test for alcohol; 12. Those who smoked more than 5 cigarettes per day on average during the 3 months prior to screening or those who do not agree to stop using any tobacco products during their stay; 13. History of surgical procedure within 3 months prior to screening or planning to undergo surgery during the study; 14. Blood donation or significant blood loss within 3 months prior to the first dose, or platelet donation within 1 month for 2 treatments. Donation of 2 therapeutic doses of platelets (1 therapeutic dose = 12 U of platelets) within 1 month; 15. Participation in a clinical trial of any drug within 3 months prior to the first dose and taking the drug; 16. Use of any drug that interacts with empagliflozin and/or CYP3A4 inducers and inhibitors , P-gp substrates , etc., within 30 days prior to the screening visit； 17. Those who have taken any prescription medication within 14 days prior to taking the medication ; 18. Anyone who has taken any over-the-counter medication, herbal medicine or health product within 7 days prior to taking the medication; 19. Those who have taken special diets (e.g. grapefruit and grapefruit-containing products), or engaged in strenuous exercise, or other factors affecting the absorption, distribution, metabolism, or excretion of the drug in the 48h prior to taking the drug; 20. Those who have consumed any xanthine-rich food 48h before taking the drug; 21. Those who have special dietary requirements and are unable to comply with the diet provided by the center and the corresponding regulations; 22. Other subjects who are judged by the investigator to be unsuitable for participation. Withdrawal Criteria and Treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 72hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-t) | 72hours
  Area under the drug concentration-time curve from time 0 to the last accurately measurable concentration at sample collection time t
Area under the plasma concentration versus time curve (AUC0-∞) | Infinite Time
  Area Under the Plasma Drug Concentration-Time Curve from Time 0 to Infinite Time
Area under the plasma concentration versus time curve (AUC0-72h) | 72hours
  Area under the drug concentration-time curve from time 0 to 72h

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University Phase I Clinical Research Center, Qingdao, Shandong, China